CLINICAL TRIAL: NCT02406664
Title: Prospective Cohort Study of the Effect of Bariatric/Metabolic Surgery on Morbid Obesity Patients With Metabolic Syndrome
Brief Title: The Effect of Bariatric/Metabolic Surgery on GFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Tae Kyung Ha, Associate Professor, Hanyang University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: NCT02271568
Record Dates: First submitted 2015-03-19; First posted 2015-04-02 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese patients (Experimental): 15 Obese patients (BMI>30) having one of comorbidity (type 2 diabetes, dyslipidemia, or hypertension) and morbid obese patients (BMI>35) accepted for bariatric surgery.
  Interventions: Procedure: Bariatric surgery
- Control patients (No Intervention): 15 matched controls receiving Intensive medical therapy

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic or Robot R-Y gastric bypass
  Arms: Obese patients

SUMMARY:
The purpose of this study is to determine the change in kidney function and blood pressure after gastric bypass versus conventional medical therapy in morbid obesity. The study mainly focus on glomerular filtration rate(GFR) with known relation to the renal function and 24 hours ambulatory blood pressure monitoring after intervention of gastric bypass or medical treatment.

DETAILED DESCRIPTION:
Metabolic syndrome is strongly associated with obesity and the patients with this syndrome are at increased risk for cardiovascular disease. Obesity constitutes a strong risk factor for the development of chronic kidney disease. Among diabetics, obesity is known to amplify the risk for kidney disease. Bariatric surgery has yielded dramatic results including longitudinal loss of excess body weight and either complete reversal or significant improvement of several features of metabolic syndrome. In addition, many observational studies have demonstrated significant reduction in proteinuria after bariatric surgery.

However, the changes in the component of cardiovascular problem among metabolic syndrome and changes in renal filtration function or progression to end stage kidney disease in morbidly obese patients after weight loss surgery have not been extensively studied. Therefore, our study mainly focus on glomerular filtration rate(GFR) with known relation to the renal function and 24 hours ambulatory blood pressure monitoring after intervention of gastric bypass or medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity (BMI>30) patients with one of comorbidity (type 2 diabetes, dyslipidemia, or hypertension)
* Morbid obese patients (BMI>35)

Exclusion Criteria:

* Prior bariatric surgery
* Malignancy (any type)
* End stage renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Glomerular filtration rate | before, 6, 12month after surgery

SECONDARY OUTCOMES:
Change in excessive body weight | before, 6, 12month after surgery
Systolic function (EF) | Before, 6 and 12month after surgery
  measured by echocardogram
Diastolic function (E,A,DT,IVRT,E/e') | Before, 6 and 12month after surgery
  measured by echocardogram
Change of daytime blood pressure (systolic blood pressure, diastolic blood pressure, mean blood pressure) | Before, 6, and 12month after surgery
  measured by 24 hours ambulatory blood pressure monitoring
Change of night time blood pressure (systolic blood pressure, diastolic blood pressure, mean blood pressure) | Before, 6, and 12month after surgery
  measured by 24 hours ambulatory blood pressure monitoring
Change of 24 hours blood pressure (systolic blood pressure, diastolic blood pressure, mean blood pressure) | Before, 6, and 12month after surgery
  measured by 24 hours ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyung Ha, MD, PhD, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Hospital, Seoul, South Korea